CLINICAL TRIAL: NCT00348023
Title: Comparison of Bimatoprost 0.03% Monotherapy vs. Dual Therapy With Travoprost 0.004% and Timolol 0.5% in Patients With Glaucoma and Ocular Hypertension
Brief Title: Bimatoprost Monotherapy vs. Dual Therapy With Travoprost and Timolol in Patients With Glaucoma and Ocular Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 5179
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2007-02-09 (Estimated); Status verified 2007-02

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Bimatoprost; Travoprost

INTERVENTIONS:
Drug: Bimatoprost 0.03%, Travoprost 0.004%, Timolol 0.5%

SUMMARY:
Evaluate the IOP-lowering efficacy and quality of life in patients using bimatoprost 0.03% monotherapy versus dual therapy with travoprost 0.004% and timolol 0.5% for the treatment of glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* · Male or female > 18 years of age

  * Diagnosis of primary open-angle glaucoma or ocular hypertension
  * Untreated IOP > 18 mm Hg in each eye at the baseline evaluation
  * Ability to provide informed consent and likely to complete all study visits

Exclusion Criteria:

* · Known contraindication to bimatoprost, travoprost, timolol, or any component of any study medication

  * Uncontrolled systemic disease
  * Active ocular disease other than POAG or ocular hypertension
  * Required use of ocular medications other than the study medications during the study (intermittent use of OTC artificial tear products will be permitted)
  * History of intraocular surgery within the last 3 months
  * Patient must not have discontinued use of any medication included in this study in the past for reasons of efficacy or intolerance

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Robert Noecker, MD, Principal Investigator — UPMC Eye Center
Locations (1):
- Dr. Noecker, Pittsburgh, Pennsylvania, United States